CLINICAL TRIAL: NCT01821599
Title: Comparative Study Between Two Physiotherapy Protocols Conventional X Accelerated in Individuals Undergoing Reconstruction of the Anterior Cruciate Ligament.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, José Carlos Alves Fabrício Júnior, Specialist, Master Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCA-9090
Record Dates: First submitted 2013-03-20; First posted 2013-04-01 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-12

CONDITIONS: Rehabilitation; Anterior Cruciate Ligament Reconstruction; Knee
Keywords: Anterior Cruciate Ligament; Knee; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional group (Active Comparator): Nonaccelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction
  Interventions: Other: Nonaccelerated Rehabilitation
- Accelerated group (Experimental): Accelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction
  Interventions: Other: Accelerated Rehabilitation

INTERVENTIONS:
Other: Nonaccelerated Rehabilitation — Nonaccelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction in 6 months of recovery.
  Arms: Conventional group
Other: Accelerated Rehabilitation — Accelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction in 4 months of recovery.
  Arms: Accelerated group

SUMMARY:
The accelerated rehabilitation and early return does not seem to be harmful, but still needs further research to define the rehabilitation time is what shows Kruse and collaborators (2012) in their study of systematic review. The surgical treatment of anterior cruciate ligament injury is the gold standard in the treatment of these injuries in young and active, the postoperative rehabilitation is extensive and full return to sport occurs only after 6 months postoperatively. Based on this gap, the investigators seek to draw properly through our study methods and more complex techniques, that comparing two rehabilitation programs can achieve high precision early rehabilitation. This will include 32 athletes who had complete ACL rupture confirmed by MRI and underwent ACL reconstruction using patellar tendon.All subjects will be followed from the pre-surgery, the fourth and sixth month after surgery with: KT1000 measures the ligamentous laxity, knee function by applying the International Knee Documentation Committee (IKDC 2000); Isokinetic Muscle Strength (Cybex). Through a random draw of sealed envelopes, patients will be allocated in their rehabilitation groups: Accelerated (4 months) or Conventional (6 months). Preoperatively, fourth and sixth month after surgery will be an assessment of laxity by (KT1000), Muscular Strength (CYBEX) and knee function affected by IKDC (2000) and Hop Test. The assessor and the patients were blinded to treatment group. This study will have the locus Institute of Orthopaedics and Traumatology, School of Medicine, São Paulo. The comparative results of the two groups are analyzed using specific statistical tests to prove an improved significative without damaging the integrity of the graft.

DETAILED DESCRIPTION:
All subjects will be followed for a period of six months. During this period will undergo three stages of evaluation.

1. º Preoperative up to two years following injury : assessment will consist KT1000 measures the ligamentous laxity, knee function by applying the International Knee Documentation Committee (IKDC 2000); Hop Test (jumps with one leg); Isokinetic Muscle Strength (Cybex).
2. º 4º months pós-surgery KT1000, International Knee Documentation Committee (IKDC 2000); Hop Test; Isokinetic Muscle Strength (Cybex)
3. º 6º months postoperatively KT1000, International Knee Documentation Committee (IKDC) + Hop Test; Isokinetic Muscle Strength (Cybex)

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of injury (primary) anterior cruciate ligament confirmed by magnetic resonance may or may not be associated with a meniscal injury or partial ligament medial collateral ligament (MCL) surgery is not indicated.
* Patients undergo surgery for anterior cruciate ligament reconstruction using patellar tendon.

Exclusion Criteria:

* Patients who had changes in diagnosis during surgery.
* Surgical complications
* Patients with More than 30% of lack or abandon physiotherapy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
KT1000 measures | Sixth months
  Measure of anterior knee stability

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC 2000) | Sixth months
  Questionnaire function subjective of the knee
Hop Test measures | sixth months
  Jump with one leg
Isokinetic of the knee measures | sixth months
  Knee Muscle Strength (Cybex).

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Fabrício, Principal Investigator — University of Sao Paulo; Roberto Mota, Study Director — University of Sao Paulo
Locations (1):
- Institute of Orthopedics and Traumatology, Faculty of Medicine of São Paulo, São Paulo, São Paulo, Brazil